CLINICAL TRIAL: NCT01967238
Title: An Open Label Study of IgG Fc Glycan Composition in Human Immunity
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TWA-0804
Record Dates: First submitted 2013-10-17; First posted 2013-10-22 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: immune response
MeSH Terms: interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Biologic/Vaccine, Age 18-64 cohort (Active Comparator): Vaccination. IM Pneumococcal, meningococcal, or flu vaccine
  Interventions: Biological: IM Pneumococcal, meningococcal, or flu vaccine
- Biologic/Vaccine, Age 65-80 cohort (Active Comparator): Vaccination. IM Pneumococcal, meningococcal, or flu vaccine
  Interventions: Biological: IM Pneumococcal, meningococcal, or flu vaccine
- Vaccine, healthy adults (Active Comparator): Vaccination. IM Pneumococcal, meningococcal, or flu vaccine
  Interventions: Biological: IM Pneumococcal, meningococcal, or flu vaccine

INTERVENTIONS:
Biological: IM Pneumococcal, meningococcal, or flu vaccine — Volunteers given one of the 3 vaccines
  Other Names: FluMist, Pneunomovax, or Menveo vaccine

SUMMARY:
In order to produce better more effective vaccines, it is important to understand the particulars of why individuals have an effective or ineffective immune response to vaccination. We are going to examine specific aspects of the antibody (IgG Fc glycan) made by healthy volunteers who receive different vaccines or who have a viral infection to understand the nature of an effective (or less effective) vaccine response. The results of this research could be used to develop adjuvants to increase/ improve vaccine response.

DETAILED DESCRIPTION:
Antibodies are principle mediators of immunity against infections and they can also give rise to autoimmune and inflammatory diseases. Two functional domains make up an IgG antibody - the Fab domain binds to a specific target, while the Fc domain can interact with receptor molecules to activate a pro- or anti- inflammatory state. The Fc domain of IgGs contains a glycan that is variable in composition and its specific sugar components are an important determinant of the biologic activity of IgGs in both protective and pathologic immune responses. New disease treatments could be developed through purposeful manipulation of IgG Fc glycans, but there is currently little known about how Fc glycan composition is regulated. We plan to study this by evaluating whether vaccination can cause changes in Fc glycan composition and, if so, whether signaling from helper T cells, age of the patient, and/or route of vaccine administration are determinants of specific modifications that are triggered by vaccination. Next, we will study effects that specific components within the Fc glycan have on immunity against the common human pathogens Streptococcus pneumoniae and influenza viruses using in vitro and in vivo models of infection. We will also study whether healthy adults who have been previously infected with dengue, zika or chikungunya virus generate distinct Fc glycoforms after vaccination compared with healthy adults who have not been previously infected with any of these viruses.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18-80 years of age
* Healthy volunteers without significant medical problems
* Able to give informed consent to participate
* Willing to receive a single dose of an FDA-approved vaccine (either the influenza virus, pneumococcal or meningococcal vaccine)
* Documented previous infection with dengue, zika or chikungunya virus or no history of dengue, zika or chikungunya infection.

Exclusion Criteria:

* Prior allergic reaction to commercial vaccination
* For Flumist participants: Close contact with person with severely compromised immune system requiring isolation
* For Flumist participants: Current illness that limits delivery to nasal airway (mild illness, such as diarrhea or mild respiratory infection with or without fever, and local infections do not apply)
* History of seizure disorder for Flumist group participants only.
* Participation in another clinical study of an investigational product currently or within the past 90 days, or expected participation during this study.
* Any clinically significant acute or chronic medical condition requiring care of a physician (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that, in the opinion of the investigator, would preclude participation.
* In the opinion of the investigator, the volunteer is unlikely to comply with the study protocol.
* Currently taking systemic steroids or other immunomodulatory medications including anticancer medications and antiviral medications.
* Egg allergy
* Received the influenza vaccine less than 1 month ago and/or received the pneumococcal and meningococcal vaccine less than 4 years ago
* Confirmed HIV infection, positive for hepatitis B surface antigen or positive for hepatitis C antibodies.
* Is pregnant or lactating
* History of Guillain-Barre syndrome
* Poor venous access
* Unable to continue participation for 12 weeks
* Any clinically significant abnormality on medical history or physical examination including history of immunodeficiency or autoimmune disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taia T Wang, MD PhD, Principal Investigator — Rockefeller Univesrity
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maamary J, Wang TT, Tan GS, Palese P, Ravetch JV. Increasing the breadth and potency of response to the seasonal influenza virus vaccine by immune complex immunization. Proc Natl Acad Sci U S A. 2017 Sep 19;114(38):10172-10177. doi: 10.1073/pnas.1707950114. Epub 2017 Sep 5. PMID 28874545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 study arms were intended, as described here.
Pre-assignment Details: 129 participants were consented; 38 were not assigned to an arm because they screened out
Period: Overall Study
Arm/Group | Biologic/Vaccine, Age 18-64 Cohort | Biologic/Vaccine, Age 65-80 Cohort | Vaccine, Healthy Adults
Started | 53 | 22 | 16
Completed | 51 | 21 | 14
Not Completed | 2 | 1 | 2
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biologic/Vaccine, Age 18-64 Cohort | Biologic/Vaccine, Age 65-80 Cohort | Vaccine, Healthy Adults | Total
Number analyzed (Participants) | 53 | 22 | 16 | 91
Age, Customized [Count of Participants; unit: Participants]
  >18 and < 65 years | 53 | 0 | 15 | 68
  >= 65 and <= 80 years | 0 | 22 | 1 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 17 | 10 | 52
  Male | 28 | 5 | 6 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 1 | 3 | 13
  Not Hispanic or Latino | 42 | 18 | 12 | 72
  Unknown or Not Reported | 2 | 3 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2 | 4
  Asian | 3 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 16 | 4 | 0 | 20
  White | 22 | 15 | 10 | 47
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 9 | 2 | 3 | 14
Region of Enrollment [Number; unit: participants]
  United States | 53 | 22 | 16 | 91

OUTCOME MEASURES:

1. Primary Outcome: The Percent (of 100%) of IgG With Galactosylation, Fucosylation and/or Sialylation
Description: The percent of Fc glycans that are galactosylation, fucosylation and/or sialylation of pre- vs. post- vaccination Fcs determined by lectin blot (Erythrina cristagalli, Aleuria Aurantia Lectin and Sambucus nigra lectins specific for galactose, fucose and 2,6-sialic acid, respectively) or by mass spectrometric analysis. 100% of IgG were found to have these modifications.
Time Frame: One Day
Population: The primary assessment in the study was intended to compare data for each Arm as shown with no comparisons by vaccine. All groups within Arm 1 were not fully enrolled, therefore it was adequately powered to perform analyses (data were not collected).
  Arm 2 was not fully enrolled and underpowered (data were not collected). Samples from Arm 3 were destroyed during the COVID-19 pandemic due to a stalled shipment which caused the samples to thaw for several days (data were not collected).
Measure: Number; unit: % of glycosylated IgG
Arm/Group | Biologic/Vaccine, Age 18-64 Cohort | Biologic/Vaccine, Age 65-80 Cohort | Vaccine, Healthy Adults
Number analyzed (Participants) | 30 | 0 | 0
% of glycosylated IgG | 100 |  |

ADVERSE EVENTS:
Time Frame: 3 years was the intended period over which each participant would be assessed. Adverse Events were monitored/assessed and collected by study cohort and not by vaccine type administered.
Groups:
- Biologic/Vaccine, Age 18-64 Cohort; Biologic/Vaccine, Age 65-80 Cohort; Vaccine, Healthy Adults: Vaccination. IM Pneumococcal, meningococcal, or flu vaccine
  IM Pneumococcal, meningococcal, or flu vaccine: Volunteers given one of the 3 vaccines
  Adverse Events were monitored/assessed and collected by study cohort and not by vaccine type administered.
Arm/Group | Biologic/Vaccine, Age 18-64 Cohort | Biologic/Vaccine, Age 65-80 Cohort | Vaccine, Healthy Adults
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/22 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/22 | 0/16
Other Adverse Events (participants affected / at risk) | 4/53 | 2/22 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biologic/Vaccine, Age 18-64 Cohort (N=53) | Biologic/Vaccine, Age 65-80 Cohort (N=22) | Vaccine, Healthy Adults (N=16)
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 0
Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Decreased white blood cell count (Immune system disorders) | 1 | 0 | 0
Shingles (Immune system disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT01967238/Prot_SAP_000.pdf
  • Informed Consent Form: Arms 1 and 2 (2016-02-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT01967238/ICF_001.pdf
  • Informed Consent Form: Arm 3 (2020-12-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT01967238/ICF_002.pdf